CLINICAL TRIAL: NCT04346641
Title: Detection of Correlation Between Facial Measurements and Tooth Size and Pulp Volume Using Cone Beam Computed Tomography
Brief Title: Correlation Between Facial Measurements and Tooth Size and Pulp Volume
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, FATMA PERTEK HATİPOĞLU, Speciality student, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: No protocol ID
Record Dates: First submitted 2020-02-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Cone-Beam Computed Tomography
Keywords: Facial measurements; Dental measurements; Cone beam computed tomography
MeSH Terms: interventions — Body Height

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Facial Measurements and Tooth Size and Pulp Volume — Radiographic images of patients who have been indicated for cone-beam computed tomography for the upper jaw for various reasons (such as impacted teeth, sinusitis, skeletal anomalies) will be reviewed retrospectively. Facial measurements (lower face height, midface height, inter-zygomatic distance, inter-pupillary distance, inter alar distance, epicanthus distance, the distance between commissures) of the patients who received cone beam computed tomography will be measured in the clinic. Mesiodistal distance, buccal palatal distance, root length, pulp volume of maxillary sixth tooth will be measured using cone beam computed tomography. The data obtained will be compared.

SUMMARY:
The aim of this study was to investigate the correlation between the measurements of the specific points of the face (lower face height, midface height, the distance between zygomatic, pupillary distance,interalar distance, epicanthus distance, the distance between commissar) and the dimensions of the maxillary sixth molar tooth (mesiodistal distance, buccal palatal distance, root length, pulp volume).

DETAILED DESCRIPTION:
Radiographic images of patients who have been indicated for cone-beam computed tomography for the upper jaw for various reasons (such as impacted teeth, sinusitis, skeletal anomalies) will be reviewed retrospectively. Facial measurements (lower face height, midface height, inter-zygomatic distance, inter-pupillary distance, interalar distance, epicanthus distance, the distance between commissures) of the patients who received cone beam computed tomography will be measured in the clinic. Mesiodistal distance, buccal palatal distance, root length, pulp volume of maxillary sixth tooth will be measured using cone beam computed tomography. The data obtained will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Upper dental arches which have maxillary first molars
* At least one tooth which has no deep caries, filling or crown restoration must be
* No resorption or pathology in the root of the tooth which disrupt integrity must be
* Healthy subjects

Exclusion Criteria:

* Deep caries, filling or crown restoration
* Resorption or pathology in the root of the tooth

Ages: 15 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Above 15 years old, healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-06-13 (Estimated); Study Completion 2020-08-13 (Estimated)

PRIMARY OUTCOMES:
Height of inferior face | 5 minute
  Distance between subnasal and gnathion
Height of medium face | 5 minute
  Distance between glabella and subnasal
bizygomatic distance | 5 minute
  Distance from the most lateral parts of the arch of the zygomas
interpupillary distance | 5 minute
  Distance the center of the pupil of the right side to the center of the pupil of the left side
interalar distance | 5 minute
  Distance from ala of one side to other
Epicanthus distance | 5 minute
  Distance from inner palpebral fissures
Commissural distance | 5 minute
  Distance from commissar of the lips
Mesiobuccal root length | 5 minute
  distance from enamel cement border of the tooth to the mesial root apex
Distobuccal root length | 5 minute
  distance from enamel cement border of the tooth to the distal root apex
Palatal root length | 5 minute
  distance from enamel cement border of the tooth to the palatal root apex
Mesiodistal width | 5 minute
  Defined as the distance between two parallel planes, tangential to the most mesial and most distal points of the crown side
Buccal palatal width | 5 minute
  Defined as the maximum distance between two parallel planes, one tangential to the most palatal point of the crown side, and the other tangential to a point on the buccal crown side
Inter first molar distance | 5 minute
  The linear distance between right and left first molar teeth between the most convex palatal crown faces
Pulp volume | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arıcıoğlu, Study Director — Recep Tayyip Erdogan University Faculty of Dentistry
Locations (1):
- Recep Tayyip Erdogan University Faculty of Dentistry, Rize, Turkey (Türkiye)